CLINICAL TRIAL: NCT05332496
Title: Efficacy and Safety of Transarterial Chemoembolization in Combination With PD-1/PD-L1 Inhibitors and Molecular Target Therapies(VEGF-TKI/Bevacizumab) for Intermediate Stage HCC
Brief Title: TACE in Combination With PD-1/PD-L1 Inhibitors and Molecular Target Therapies for Intermediate HCC
Acronym: CHANCE2202
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: CHANCE2202
Record Dates: First submitted 2022-04-02; First posted 2022-04-18 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; transarterial chemoembolization; immune checkpoint inhibitors; molecular target therapies; Intermediate stage
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: TACE+PD-1/PD-L1 inhibitors+VEGF-TKI/bevacizumab: TACE was performed up to 3 months after the first PD-1/PD-L1 inhibitor/anti-angiogenic drug treatment or within 1 month before treatment. The interval between first use PD-1/PD-L1 inhibitors and anti-angiogenesis drugs ≤1 week；
  Interventions: Drug: PD-1/PD-L1 inhibitors+VEGF-TKI/bevacizumab; Procedure: TACE
- Control group: TACE: TACE monotherapy
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: PD-1/PD-L1 inhibitors+VEGF-TKI/bevacizumab — PD-1/PD-L1 inhibitors: atezolizumab, sintilimab, pembrolizumab, nivolumab, camrelizumab, tislelizumab, toripalimab, durvalumab, penpulimab, and other ICIs; VEGF-TKI/bevacizumab: sorafenib, lenvatinib, donafenib, apatinib, anlotinib, bevacizumab/ bevacizumab biosimilar, and other anti-angiogenesis drugs; Both PD-1/PD-L1 inhibitors and anti-angiogenesis drugs only include marketed drugs but are not limited to HCC approval.
  Groups: Study group: TACE+PD-1/PD-L1 inhibitors+VEGF-TKI/bevacizumab
Procedure: TACE — TACE: cTACE (conventional TACE) or dTACE (drug-eluting beads TACE);

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of transarterial chemoembolization (TACE) in combination with PD-1/PD-L1 Inhibitors and molecular target therapies in patients with Intermediate-stage hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) can induce immunogenic cell death and tumor-specific immune response which results in the release of tumor antigens and transform "cold" tumors with lacking immune effector cells into "hot" tumors with immune effector cells infiltration. This provides a theoretical basis for TACE combined with immune checkpoint inhibitors (ICIs) in hepatocellular carcinoma (HCC) patients. The purpose of this study is to evaluate the safety and efficacy of transarterial chemoembolization (TACE) in combination with PD-1/PD-L1 Inhibitors and molecular target therapies(including, VEGF-TKI/ bevacizumab) in patients with Intermediate-stage HCC. This real-world study also would like to explore the optimal combined treatment and subgroup of HCC patients for providing further information for clinical practice and trials.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Barcelona Clinic Liver Cancer (BCLC) stage B, without the presence of extrahepatic spread and/or macrovascular invasion;
3. Has not received any previous TACE/HAIC and systemic therapy for HCC (including chemotherapy, molecularly targeted therapy, immunotherapy);
4. Both PD-1/PD-L1 inhibitors and anti-angiogenesis drugs patients received only include marketed drugs but are not limited to HCC approval;
5. TACE was performed after the first PD-1/PD-L1 inhibitor/anti-angiogenic drug treatment or before treatment;
6. Received at least 1 cycle of PD-1/PD-L1 inhibitor/anti-angiogenic drug combination therapy after TACE treatment；
7. Has repeated measurable intrahepatic lesions according to mRECIST;

Exclusion Criteria:

1. Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes(confirmed by histology, or pathology) are not eligible;
2. Unable to meet criteria of combination timeframe described above;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate HCC who received TACE in combination with PD-1/PD-L1 inhibitors and molecular target therapies under real-world practice conditions.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.
Overall Survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
PFS per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to RECIST 1.1) or death due to any cause, whichever occurs first.
Objective response rate(ORR) per mRECIST | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per mRECIST.
Duration of Response (DOR) per mRECIST | up to approximately 2 years
  DOR is determined by disease assessment and is defined as the time from the first documented evidence of a response of CR or PR until the first documented disease progression (according to mRECIST) or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) per mRECIST | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD) per mRECIST.
ORR per RESCIST 1.1 | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
DOR per RESCIST 1.1 | up to approximately 2 years
  DOR is determined by disease assessment and is defined as the time from the first documented evidence of a response of CR or PR until the first documented disease progression (according to RESCIST 1.1) or death due to any cause, whichever occurs first.
DCR per RESCIST 1.1 | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD)per RESCIST 1.1.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D., Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China; Zheng-Gang Ren, M.D., Principal Investigator — Liver Cancer Institute, Zhongshan Hospital, Fudan University, Shanghai, China
Locations (2):
- China (2):
  - Gao-Jun Teng, Nanjing
  - Zheng-Gang Ren, Nanjing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llovet JM, Villanueva A, Marrero JA, Schwartz M, Meyer T, Galle PR, Lencioni R, Greten TF, Kudo M, Mandrekar SJ, Zhu AX, Finn RS, Roberts LR; AASLD Panel of Experts on Trial Design in HCC. Trial Design and Endpoints in Hepatocellular Carcinoma: AASLD Consensus Conference. Hepatology. 2021 Jan;73 Suppl 1:158-191. doi: 10.1002/hep.31327. Epub 2020 Sep 9. No abstract available. PMID 32430997
- [Background] Llovet JM, Kelley RK, Villanueva A, Singal AG, Pikarsky E, Roayaie S, Lencioni R, Koike K, Zucman-Rossi J, Finn RS. Hepatocellular carcinoma. Nat Rev Dis Primers. 2021 Jan 21;7(1):6. doi: 10.1038/s41572-020-00240-3. PMID 33479224
- [Background] Ochoa de Olza M, Navarro Rodrigo B, Zimmermann S, Coukos G. Turning up the heat on non-immunoreactive tumours: opportunities for clinical development. Lancet Oncol. 2020 Sep;21(9):e419-e430. doi: 10.1016/S1470-2045(20)30234-5. PMID 32888471
- [Background] Pinato DJ, Murray SM, Forner A, Kaneko T, Fessas P, Toniutto P, Minguez B, Cacciato V, Avellini C, Diaz A, Boyton RJ, Altmann DM, Goldin RD, Akarca AU, Marafioti T, Mauri FA, Casagrande E, Grillo F, Giannini E, Bhoori S, Mazzaferro V. Trans-arterial chemoembolization as a loco-regional inducer of immunogenic cell death in hepatocellular carcinoma: implications for immunotherapy. J Immunother Cancer. 2021 Sep;9(9):e003311. doi: 10.1136/jitc-2021-003311. PMID 34593621